CLINICAL TRIAL: NCT01175512
Title: Novel Interventions to Reduce Stress Induced Non-homeostatic Eating
Brief Title: Stress, Hormones, and Eating
Acronym: SHE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 1U01HL097973-01 (NIH)
Record Dates: First submitted 2010-07-28; First posted 2010-08-04 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Food Addiction; How Opioid Tone Was Related to Self Reported; Drive to Eat Using a Measure of Food Addiction
Keywords: naltrexone; obesity; cortisol; food addiction
MeSH Terms: conditions — Food Addiction; Obesity | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Naltrexone (Active Comparator): 4 days, counterbalanced dosing of 25mg, 50mg, placebo, placebo.
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator): 4 days, counterbalanced dosing of 25mg, 50mg, placebo, placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — 4 days, counterbalanced dosing of 25mg, 50mg, placebo, placebo.
  Arms: Naltrexone
Drug: Placebo — 4 days, counterbalanced dosing of 25mg, 50mg, placebo, placebo.
  Arms: Placebo

SUMMARY:
The investigators will develop a measure of endogenous opioid tone that might serve as a biological marker for drive for palatable food. Using a 'naltrexone probe,' the investigators will assess whether individual response to one dose of an opioid receptor antagonist, naltrexone, is related to non-homeostatic eating in non-pregnant women.

Hypothesis 1: Naltrexone Response will be related to non-homeostatic eating.

Hypothesis 2: Response profiles to the 25 mg dose will be slightly less in magnitude than the 50 mg dose. However, responses will be similarly related to non-homeostatic eating measures.

Hypothesis 3: Response to naltrexone will be highly stable within individuals across time, in the absence of an intervention.

DETAILED DESCRIPTION:
Opioid tone may provide a way to identify people at risk of reward based eating, with more accuracy than self-report measures. Knowing such risk could improve treatment matching, and provide a biomarker to assess treatment progress. There is no direct measure of central opioid activity in humans, short of PET scans for opioid receptor binding. However, there is a promising indicator using an opioid antagonist such as naltrexone. Blocking opioid receptor releases the inhibitory opioidergic inputs to hypothalamic corticotropic releasing hormone (CRH) neurons, thus increasing CRH, and eventually cortisol in the blood. The extent of the cortisol rise in response to naltrexone might serve as an indicator of endogenous opioidergic tone. It is hypothesized that greater increases in cortisol indicate weaker endogenous opioid activity (by indicating a more complete opioid blockade). Salivary cortisol response to naltrexone may offer a relatively safe and unobtrusive way to measure endogenous opioidergic tone. We propose to test the reliability and validity of the naltrexone probe, taken at home, as a measure of endogenous opioidergic tone. In a previous study (Daubenmier et al, 2013), we administered a one time 50mg dose of naltrexone and examined nausea and cortisol responses. Results suggested that responses were higher in those who showed greater drive to eat. Here we examine a more direct measure of drive to eat, using the Yale Food Addiction Scale (YFAS), and test whether nausea and cortisol responses were associated with greater drive to eat, whether 50mg produced greater responses than 25 mg, and whether the responses were stable (highly related) when tested again one month later.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age > 20 to 45 years (pre-menopausal women)
* BMI > 30 and no larger than BMI = 40 or 300 pounds

Exclusion Criteria:

* Inability to provide informed consent or speak English
* Needle phobic or fainting in response to blood draw
* Diabetes
* Currently pregnant or breastfeeding
* Currently Smoke
* Bulimia (Binge Eating Disorder is common among the obese, and allowed)
* Pacemaker
* Shift Worker
* Beta Blocker Medication use
* Liver Medication use
* Weight Loss Medication use
* Chronic current use of cortisol containing medications
* Kidney Disease (based on elevated Blood Urea Nitrogen and Creatinine)
* Illegal Drug Use (presence in urine)
* Liver Cirrhosis or Acute hepatitis (based on elevated Alanine transaminase)
* Substance abuse, mental health, or medical condition that, in the opinion of investigators, will affect study outcomes (e.g., hypertension, severe food allergies).

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Ideal Dosage | May 2012
  1) To examine criterion validity by testing whether level of opioid tone (based on response to naltrexone probe) is associated with self reported scores on non-homeostatic eating measures, behavioral and cognitive tasks assessing constructs related to addiction (eg, impulsivity) and ideal dosage (25 vs. 50 mg) in 60 obese women.

SECONDARY OUTCOMES:
Test Retest Reliability | May 2012
  2) To examine test-retest reliability of naltrexone response one month later
Home Based Measures Reliability | May 2012
  3) To examine the reliability of home based measures. In other words, we will test whether cortisol and nausea responses taken in clinic, which are taken at highly controlled (accurate) times, are comparable to the responses from samples taken at home using saliva measures.

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Epel, PhD, Principal Investigator — University of California, San Francisco

REFERENCES:
- [Background] Gearhardt AN, Corbin WR, Brownell KD. Preliminary validation of the Yale Food Addiction Scale. Appetite. 2009 Apr;52(2):430-6. doi: 10.1016/j.appet.2008.12.003. Epub 2008 Dec 11. PMID 19121351
- [Background] Daubenmier J, Lustig RH, Hecht FM, Kristeller J, Woolley J, Adam T, Dallman M, Epel E. A new biomarker of hedonic eating? A preliminary investigation of cortisol and nausea responses to acute opioid blockade. Appetite. 2014 Mar;74:92-100. doi: 10.1016/j.appet.2013.11.014. Epub 2013 Nov 27. PMID 24291355